CLINICAL TRIAL: NCT03586700
Title: Based on the Ultrasound Evaluating the Effect of Xiaozhong Fang Particles for Knee Osteoarthritic With Synovial Fluid
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, mei han, Assistant Researcher, Beijing University of Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: QN2016-03
Record Dates: First submitted 2018-05-25; First posted 2018-07-16 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; Synovium effusion; RCT; placebo
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xiao zhong fang granules (Experimental): Xiao zhong fang granules were made from Smilax glabra 20g, Paris polyphylla 10g, Alisma orientale15g, Plantago15g, Peach kernel 10g, safflower 10g, radices cyathulae10g,fructus chaenomeles lagenaria 10g, corydalis tuber 10g, radix clematis 10g, radices paeoniae alba 10g, glycyrrhiza 10g. Granules 6 days for one course, continuously taking two courses, interval of 1 day, and then take 2 courses. Short wave infrared radiation treatment every other day, ensure 3 times in 7 days, 7 days for a course of treatment, continuously for 4 courses.
  Interventions: Drug: Xiao zhong fang granules; Radiation: Short wave infrared radiation
- Placebo Xiao zhong fang granules (Placebo Comparator): Placebo Xiao zhong fang granules were made by the same institution. Placebo granules 6 days for one course, continuously taking two courses, interval of 1 day, and then take 2 courses. Short wave infrared radiation treatment every other day, ensure 3 times in 7 days, 7 days for a course of treatment, continuously for 4 courses.
  Interventions: Radiation: Short wave infrared radiation; Drug: Placebo Xiao zhong fang granules

INTERVENTIONS:
Drug: Xiao zhong fang granules — Chinese medicine Xiao zhong fang was Professor Sun Chengxiang's experience formula in Massage Department of Dongzhimen Hospital. The function of the formula is to activate blood circulation and dredge collaterals, tonifying kidney and promoting dampness to soothe the liver and nourish tendons.
  Arms: Xiao zhong fang granules
Radiation: Short wave infrared radiation — Short waves infrared radiation treatment every other day, ensure 3 times in 7 days, 7 days for a course of treatment, continuously for 4 courses.
Drug: Placebo Xiao zhong fang granules — Made of starch,dextrin and edible pigment from Dongzhimen Hospital of Beijing university of chinese medicine.
  Arms: Placebo Xiao zhong fang granules

SUMMARY:
This study is a randomized, single blind, controlled trial. Aim to compare the effectiveness (especially the absorption degree of the synovial effusion measured by B ultrasonic) of the treatment group with the control group. The treatment group was given Xiao zhong fang granules orally and short wave infrared radiation and the control group was given the placebo Xiao zhong fang granules orally and short wave infrared radiation. To evaluate the clinical efficacy of the Chinese medicine in the treatment of the synovial effusion of knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* 1) the American Society of Rheumatology established the diagnostic criteria for knee OA in 2001;
* 2) Kellgren/Lawrence score of knee joint grade as I,II and early III.
* 3) According to "Principles of clinical guidance for new drugs of traditional Chinese Medicine ",diagnosed as "Xi Bi Disease".
* 4) Patients with informed consent.
* 5)Blood and urine routine tests, liver and kidney functions, electrocardiogram were normal before recruitment.
* 6) Patients were not treated with NSAIDS drugs or hormone drugs, and no patients were treated with drugs related to this disease at least 2 weeks.

Exclusion Criteria:

* 1)Patients suffer from other rheumatic and metabolic diseases such as gout, rheumatoid arthritis, diabetes and so on.
* 2) Patients with knee joint inflammatory infection, such as suppurative and nonspecific.
* 3)Patients accompanied by traumatic synovitis, Villonodular pigmented synovitis, synovial membrane of the knee is the main lesion.
* 4) Patients with informed consent.
* 5)The color of joint fluid of patients' knees is pink or other color or cloudy; the white blood cell counts > 1000 /mm3 or with crystal in the joint fluid.
* 6)Patients blood RF > 30IU/ml, ESR > 20mm/h, CRP > 10mg/L.
* 7)Patients combined with severe cardiovascular, cerebrovascular, liver, kidney and other primary diseases and mental diseases.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-09-15 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Walther grading of synovial effusion of Knee joint | After treatment(28days)
  The Walther grading standard of the synovial effusion of the knee joint (measuring the anterior and posterior diameter of the effusion): the 0 level is the joint cavity without effusion or the expansion of joint capsule<2mm; the grade I is a small amount of effusion, the expansion of joint capsule is 2mm-5mm; the grade II is a medium amount of effusion, the expansion of joint capsule is 6mm-10mm; the grade III is a large amount of effusion, and the joint capsule expands >10mm.

CONTACTS AND LOCATIONS:
Overall Officials: DUODUO LI, MASTER, Principal Investigator — Dongzhimen Hospital, Beijing
Locations (1):
- Dongzhimen Hospital Beijing University of Chinese Medicine, Beijing, Bejiing, China

IPD SHARING:
Plan to Share IPD: Undecided